CLINICAL TRIAL: NCT05543369
Title: A Phase I, Single-Centre, Open-Label, Repeat Dose Study to Assess the Pharmacokinetics, Safety and Tolerability Following Administration of Elafibranor in Healthy Japanese and Non-Asian Participants.
Brief Title: Study to Compare the Level of Elafibranor in Blood After Repeat Administration in Japanese and Non-Asian Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLIN-60190-450
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Elafibranor
MeSH Terms: interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 : Healthy Japanese Participants (Experimental): Participants will receive Elafibranor 80 mg once daily on Day 1 to Day 18.
  Interventions: Drug: Elafibranor
- Cohort 2: Healthy Non-Asian Participants (Experimental): Participants will receive Elafibranor 80 mg once daily on Day 1 to Day 18.
  Interventions: Drug: Elafibranor

INTERVENTIONS:
Drug: Elafibranor — Oral Tablet
  Other Names: GFT505

SUMMARY:
This study is intended to measure the blood levels of Elafibranor and one of its metabolites in Japanese and non-Asian Healthy Participants, to be able to compare how the body absorbs, distributes, and eliminates Elafibranor after Repeat Administration, in order to support inclusion of Japanese patients in the planned clinical studies with elafibranor.

ELIGIBILITY:
Inclusion Criteria :

* Participants should meet one of the following ethnicity criteria:

  1. Japanese:

     * Must have been born in Japan.
     * Both the subject's biological parents and all four biological grandparents must be Japanese, as confirmed by interview.
     * Must not be living outside of Japan for more than 10 years.
     * Lifestyle, including diet, has not changed significantly since leaving Japan
  2. Non-Asian:

     * Must be a descent from North America, South America, Europe or the Middle East (subjects from Asian/Pacific Islander and African American descent are excluded).
     * Both the subject's biological parents and all four biological grandparents must be of non-Asian descent
* Male or female participants must be 18 to 55 years of age (inclusive) at the time of signing the informed consent. A minimum of six evaluable subjects of each sex will have to be completed within each cohort (i.e. at least six female and six male subjects)
* Has provided signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Willingness to remain at the clinic for the required duration and willingness to return to the clinic for the follow-up evaluation as specified in the protocol
* Healthy participants as determined by medical evaluation at the screening visit including medical history, physical examination, laboratory tests, electrocardiogram (ECG) and vital signs monitoring
* Laboratory parameters within the normal range of the laboratory (haematological, blood biochemistry, urinalysis). Individual values out of the normal range can be accepted if judged non-clinically significant by the investigator.
* Normal ECG recording on a 12-lead ECG at screening and at admission (Day -1):

  * 120≤PR≤220 ms,
  * QRS<110 ms,
  * QTcF≤430 ms for male and ≤450 ms for female,
* No evidence of sinus node automaticity or abnormal conduction, or rhythm disorders of concern, except as considered non-clinically significant by the investigator. Out-of-range values that are not clinically significant (as determined by the investigator) may be repeated twice during screening and admission and the participant may be enrolled if at least one repeated value is within the range noted above.
* Normal blood pressure (BP) and heart rate (HR) at the screening and at admission after 5 minutes in supine position:

  * 90 mmHg ≤ systolic blood pressure (SBP)≤145 mmHg
  * 50 mmHg ≤ diastolic blood pressure (DBP)≤90 mmHg,
  * 45 bpm≤HR≤90 bpm,
* For these parameters, out-of-range values that are not clinically significant (as determined by the investigator) may be repeated twice during screening and admission and the participant may be enrolled if at least one repeated value is within the range noted above.
* Body weight not below 45 kg and body mass index (BMI) within the range 18.0 kg/m^2 and 30.0 kg/m^2
* Contraception/Barrier Requirements:

  1. Female participants:

     * A female participant is eligible to participate if she is not pregnant or breastfeeding at screening, is willing not to become pregnant during the study and one of the following conditions applies:
     * Is a woman of nonchildbearing potential (WONCBP), or
     * Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the study intervention period and for at least one month after the last dose of study intervention. The investigator should evaluate the potential for contraceptive method failure (e.g. noncompliance, recently initiated) in relationship to the first dose of study intervention.
     * A WOCBP must have a negative highly sensitive pregnancy test (serum as required by local regulations) within 24 hours before dosing with study intervention. The investigator is responsible for review of medical history, menstrual history and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
  2. Male participants:

     * Male participants are eligible to participate if they agree to the following during the intervention period and for at least 90 days after the last dose of study intervention:
     * Refrain from donating sperm PLUS, either:
     * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, or
     * Must agree to use contraception /barrier as detailed below:
     * Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak and there remains a risk to pregnant women and women of childbearing potential

Exclusion Criteria :

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, haematological or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Lymphoma, leukaemia or any malignancy within the past 5 years except basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years prior to screening
* Breast cancer within the past 10 years prior to screening
* Major surgery within 28 days prior to screening
* History of COVID-19 infection (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated) within 2 months before dosing
* Past or intended use of over the counter (OTC) or prescription medication (including herbal medications or vitamin supplements, nutritional supplements, herb-containing drug preparations (including Chinese medicines) within 14 days (or 5 half-lives of the drug (whichever is longer) prior to dosing. Exceptions are oral contraception/hormone replacement therapy for females and paracetamol/acetaminophen at doses of ≤2 g/day
* Any vaccination during the 4 weeks before enrolment or planned during the clinical study
* Use of any medications within 3 months that may interfere with absorption, distribution, metabolism or excretion of the study intervention, or any medication that may result in induction or inhibition of microsomal enzymes
* Plasma donation within 14 days of the screening or any blood donation/blood loss >450 mL during the last 30 days before screening. Blood and/or plasma should not be donated until 30 days after last study intervention
* Current enrolment or past participation within the last 3 months (or 5 half-lives, whichever is longer) before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research
* Presence of hepatitis B surface antigen (HBsAg) at screening
* Positive hepatitis C antibody test result at screening. NOTE: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled if a confirmatory negative hepatitis C ribonucleic acid (RNA) test is obtained and sustained viral response can be documented
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention. NOTE: Test is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing
* Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) Polymerase chain reaction (PCR) test result at screening or admission
* Positive drugs of abuse/alcohol screen at screening and at admission
* Positive human immunodeficiency virus (HIV) antibody test at screening
* Consumption of other foods or beverages (red wine, Seville oranges, grapefruit or grapefruit juice (including pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices)) that may affect drug-metabolising enzymes or transporters from 7 days prior to dosing until discharge
* History of drug or alcohol abuse or excessive intake of alcohol within the 12 months prior to first dosing, or evidence of such abuse as indicated by the laboratory assays conducted at screening or admission. Intake of alcohol above the official recommendation, defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for women. Inability to abstain from alcohol for 24 hours before dosing until discharge
* Inability to abstain from ingesting caffeine- or xanthine containing products (e.g. coffee, tea, cola drinks, energy drinks and chocolate) for 24 hours before dosing until discharge
* History of illicit drug abuse within the last 12 months
* Sensitivity to any components of the study intervention or other allergy that, in the opinion of the investigator, contraindicates participation in the study, including lactose intolerance
* Inability to abstain from intensive muscular effort. Participants should not engage in any strenuous activity from 72 hours prior to admission to the CRU until after their discharge
* Smoking or use of tobacco or nicotine-containing products (including nicotine patches) within 3 months prior to dosing, during the study until discharge. Status will be confirmed with a urine cotinine at screening and at admission
* Had been on a diet incompatible with the on-study diet (i.e. unusual meal habits, special diet requirements or unwillingness to eat the food provided in the study, e.g. vegetarian nor vegan), in the opinion of the investigator or designee, within the 30 days prior to the first dosing and throughout the study
* Venous status at forearm or dorsal hand making it difficult to insert a venous peripheral catheter
* Vulnerable subjects, e.g. kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Noncompartmental Pharmacokinetics (PK) of Elafibranor and its Metabolite GFT1007: Area Under the Concentration-time Curve Over the Dosing Interval from Time 0 to 24 hours(AUCτ) | Day 1 and Day 18
  AUCτ will be recorded from the PK blood samples collected.
Noncompartmental PK of Elafibranor and its Metabolite GFT1007: Maximum (peak) Observed Plasma Drug Concentration (Cmax) | Day 1 and Day 18
  Cmax will be recorded from the PK blood samples collected.
Noncompartmental PK of Elafibranor and its Metabolite GFT1007: Time to Maximum Observed Drug Concentration (Tmax) | Day 1 and Day 18
  Tmax will be recorded from the PK blood samples collected.
Noncompartmental PK of Elafibranor and its Metabolite GFT1007: Trough Observed Plasma Concentration Before Dosing or at the end of the Dosing Interval (Ctrough) | Day 1 and Day 18
  Ctrough will be recorded from the PK blood samples collected.
Geometric Mean Ratios (GMR) of Elafibranor and and its Metabolite GFT1007: Area Under the Concentration-time Curve Over the Dosing Interval from Time 0 to 24 hours(AUCτ) at Steady State | Day 18
  AUCτ at steady state will be recorded from the PK blood samples collected.
GMR of Elafibranor and and its Metabolite GFT1007: Maximum (peak) Observed Plasma Drug Concentration (Cmax) at Steady State | Day 18
  Cmax at steady state will be recorded from the PK blood samples collected.

SECONDARY OUTCOMES:
Percentage of Participants With Clinically Significant changes in Laboratory Parameters (blood chemistry, hematology and coagulation) | Baseline up to Day 19
  Percentage of participants with clinically significant change in laboratory parameters (blood chemistry, hematology and coagulation) will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Clinically Significant Changes in Physical Examination | Baseline up to Day 19
  Percentage of participants with clinically significant changes in physical examination findings will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Readings | Baseline up to Day 19
  Percentage of participants with clinically significant changes in ECG readings will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Clinically Significant Changes in Vital Signs | Baseline up to Day 19
  Percentage of participants with clinically significant changes in Vital Signs will be reported. The clinical significance will be decided by the investigator.
Percentage of Participants With Treatment Emergent Adverse Event (TEAEs) and Adverse Events of Special Interest (AESIs) | Baseline up to Day 19
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- United States (2):
  - Collaborative Neuroscience Research LLC, Long Beach, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2024/03/15152815/LaySummary_Phase_I_Study_of_Elafibranor_in_Healthy_Asian_Volunteers_715537_01_March_2024.pdf